CLINICAL TRIAL: NCT01910727
Title: Together on Diabetes Study: Evaluation of a Pilot Diabetes Prevention and Management Program for American Indian Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Together on Diabetes - JHSPH
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Diabetes
Keywords: American Indian; Diabetes; Pre-diabetes; Family health Coach
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Together on Diabetes-Hopkins (Experimental)
  Interventions: Behavioral: Together on Diabetes-Hopkins

INTERVENTIONS:
Behavioral: Together on Diabetes-Hopkins — The Johns Hopkins Center for American Indian Health, with support from Bristol-Myers Squibb Foundation, Inc. is adapting a Family Health Coach model for diabetes prevention with four southwestern tribal communities. Specifically, Johns Hopkins Center for American Indian Health has designed a paraprofessional delivered pilot intervention aimed at improving the prevention and management of type 2 diabetes among American Indian youth. For Youth Participants, the pilot intervention consists of 12 sessions delivered during a 6-month intervention phase, plus 6 check-ins delivered during a 6-month follow-up phase. For Support Persons, the pilot intervention consists of 4 family skill building sessions delivered during the first 4 months of the Youth Participant's intervention phase.

SUMMARY:
The objective of the Together on Diabetes study is to test the efficacy of a pilot intervention to improve the prevention and management of type 2 diabetes among American Indian youth.

The primary aim of this study is to determine the impact of the Together on Diabetes pilot intervention on youth diabetes risk behaviors, including:

* Improvement in youth dietary intake, with a specific focus on reducing the percent of total calories from fat.
* Improvement in youth physical activity, with a specific focus on increasing the number of minutes of physical activity each week.

An additional primary aim of the study is to determine the feasibility and acceptability of the pilot intervention and evaluation, including program adherence and program satisfaction.

The secondary aim of this study is to determine the feasibility of collecting data to determine program impact on a number of physiological measures.

DETAILED DESCRIPTION:
This is a single group pre-post study designed to evaluate the feasibility and effectiveness of a pilot intervention at improving the prevention and management of type 2 diabetes among American Indian youth. The intervention uses a Family Health Coach model to work with families of youth with diabetes or at high risk of diabetes. Health Coaches visit families in their homes and conduct intervention sessions with both youth and a designated adult 'support person' (e.g., parent, guardian, etc). For Youth Participants, the pilot intervention consists of 12 sessions (45-60 minutes in duration) delivered during a 6-month intervention phase, plus 6 check-ins delivered during a 6-month follow-up phase. There are also 4 optional social support visits for the Youth Participants in order to provide necessary assistance with challenges the youth may be facing. For Support Persons, the pilot intervention consists of 4 family skill building sessions (20-30 minutes in length) delivered during the first 4 months of the Youth Participant's intervention phase. Support Persons will also be welcomed and encouraged to attend any of the Youth Participant sessions. All sessions are designed to be taught at the participant's home, but they may also occur at another location chosen by the participant (e.g. school, study office, clinic). Outcome data will be collected at Baseline, 3 months following Baseline, 6 months following Baseline, and 12 months following Baseline.

ELIGIBILITY:
Inclusion Criteria:

(YOUTH PARTICIPANT) --

* American Indian youth aged 10-19 years old at enrollment
* Resides within 1-hour transportation range (~ 50 miles) of the participating Indian Health Service (IHS) medical facilities (Tuba City, Arizona; Chinle, Arizona; Shiprock, New Mexico; Whiteriver, Arizona).
* Parent/guardian consent for youth under 18 years old.
* Referral from an Indian Health Services provider indicating a diagnosis by laboratory test of type 2 diabetes or pre-diabetes OR considered at-risk for type 2 diabetes based on BMI ≥ 85th percentile and qualifying lab test

(SUPPORT PERSON) --

* Adults 18 years of age or older
* Identified on the Youth Participant consent form as the preferred Support Person to be enrolled in the program
* Living with the enrolled Youth Participant or within 15 miles of the youth

Exclusion Criteria:

(YOUTH PARTICIPANT)

* Females who are pregnant or nursing or are planning to become pregnant within one year of enrollment
* Diabetes due to secondary causes, such as exogenous steroids, Cushing's, or Cystic Fibrosis
* Youth with type 1 diabetes.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 506 (Actual)
Dates: Start 2011-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in percent of total calories from fat from baseline through 12 months follow-up | 12 months follow-up

SECONDARY OUTCOMES:
Increased physical activity levels between baseline and 12 months follow-up | 12 months follow-up
Decreased body mass index between baseline and 12 months follow-up | 12 months follow-up
Improvement in point of care Hemoglobin A1C level between baseline and 12 month follow-up | 12 months follow-up
Decrease in waist circumference between baseline and 12 months follow-up | 12 months follow-up
Decreased blood pressure between baseline and 12 months follow-up | 12 months follow-up
Improvements in youth diabetes knowledge test score between baseline and 12 months follow-up | 12 months follow-up
Improved score on Pediatric quality of life assessment (Ped-QL) between baseline and 12 months follow-up | 12 months follow-up
Increased numbers of family members involved in diabetes support care between baseline and 12 months follow-up | 12 months follow-up
Increased numbers of individuals having been screen for diabetes between baseline and 12 months follow-up | 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, MPH, MA, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No